CLINICAL TRIAL: NCT00266552
Title: The Safety And Efficacy Of Risperidone Versus Placebo In Conduct Disorder and Other Disruptive Behavior Disorders In Mild, Moderate And Borderline Mentally Retarded Children Aged 5 To 12 Years
Brief Title: A Study of the Safety and Effectiveness of Risperidone Versus Placebo for the Treatment of Conduct Disorder in Children With Mild, Moderate, or Borderline Mental Retardation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006019
Record Dates: First submitted 2005-12-16; First posted 2005-12-19 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Conduct Disorder; Disruptive Behavior Disorder; Oppositional Defiant Disorder
Keywords: conduct disorder; oppositional defiant disorder; disruptive behavior disorder not otherwise specified; ADHD; risperidone; antipsychotropic agents; children
MeSH Terms: conditions — Conduct Disorder; Attention Deficit and Disruptive Behavior Disorders; Oppositional Defiant Disorder; Attention Deficit Disorder with Hyperactivity | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of the study is to assess the effectiveness and safety of an oral solution of risperidone (an antipsychotic medication) versus placebo in the treatment of conduct disorder in children with mild, moderate, or borderline mental retardation.

DETAILED DESCRIPTION:
Conduct and psychiatric disorders are found among a higher proportion of people with mental retardation than among people who are not mentally retarded. Among the many different treatment approaches to conduct disorder are drug therapy, behavioral treatment, psychotherapy, and training for cognitive and social skills. Studies have suggested that neuroleptic drugs, such as risperidone, may be beneficial in treating conduct disorder in mental retardation. This is a randomized, double-blind, placebo-controlled study to evaluate the effectiveness of risperidone (0.02 to 0.06 mg/kg/day) compared with placebo in the treatment of children 5 to 12 years of age with mild, moderate, or borderline mental retardation, and who display destructive behaviors. The study has two phases: a run-in phase of 1 week and a treatment phase of 6 weeks. Patients receive placebo to be taken orally once a day during the first week (run-in). On the basis of scores on the Nisonger Child Behavior Rating Form (N-CBRF) and the Vineland Adaptive Behavior Scale after the first week, patients either continue in the double-blind treatment phase or discontinue the study. During the treatment phase patients receive an oral solution of risperidone (increasing gradually to a maximum dose of 0.06 mg/kg) or placebo to be taken once daily for 6 weeks. A parent or caregiver evaluates the child's behavior and symptoms at scheduled office visits during the course of treatment. The primary measure of effectiveness is the change in the Conduct Problem subscale of the Nisonger Child Behavior Rating Form (N-CBRF) at end of treatment compared with baseline. Additional assessments of effectiveness include: the Aberrant Behavior Checklist (ABC), the Behavioral Problems Inventory (BPI), and the Clinical Global Impression (CGI). Safety assessments include the incidence of adverse events throughout the study; weekly measurement of vital signs (pulse, temperature, blood pressure) and evaluation of the presence and severity of extrapyramidal symptoms by the Extrapyramidal Symptom Rating Scale (ESRS); and clinical laboratory tests performed both before study initiation and at the end of treatment. The study hypothesis is that risperidone is well tolerated and effective for the treatment of conduct disorder in children aged 5 to 12 years with mild, moderate, or borderline mental retardation. Risperidone oral solution 1 mg/mL or placebo oral solution, once daily on Days 1 and 2 at dose of 0.01 mg/kg body weight. Dose is 0.02 mg/kg on Day 3, increasing gradually to 0.06 mg/kg (maximum) once daily through 6 weeks. Dosage may be increased or decreased at investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Conduct Disorder, Oppositional Defiant Disorder, or Disruptive Behavior Disorder not otherwise specified, by the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV), Axis I criteria (patients with conduct disorder who also meet DSM-IV criteria for Attention Deficit/Hyperactivity Disorder (AD/HD) are eligible)
* total rating of >=24 on the Nisonger Child Behavior Rating Form (N-CBRF) Conduct Problem Subscale
* Diagnosis of Mild Mental Retardation, Moderate Mental Retardation or Borderline Intellectual Functioning by DSM-IV Axis II criteria (represents intelligence quotients (IQs) ranging from 35 to 84)
* Vineland Adaptive Behavior Scale <=84.

Exclusion Criteria:

* Diagnosis of Pervasive Development Disorder or Schizophrenia and/or Other Psychotic Disorders by DSM-IV criteria
* mental impairment caused by head injury
* seizure disorder currently requiring medication
* history of tardive dyskinesia (a complication of neuroleptic therapy involving involuntary movements of facial muscles) or neuroleptic malignant syndrome (a rare psychotropic-drug reaction, which may be characterized by confusion, reduced consciousness, high fever or pronounced muscle stiffness)
* known hypersensitivity, intolerance, or unresponsiveness to risperidone.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Study Completion 1998-10 (Actual)

PRIMARY OUTCOMES:
Change in the Conduct Problem subscale of the Nisonger Child Behavior Rating Form (N-CBRF) at end of treatment compared with baseline

SECONDARY OUTCOMES:
Changes in Aberrant Behavior Checklist (ABC), Behavioral Problems Inventory (BPI), and Clinical Global Impression (CGI) at end of treatment compared with baseline; incidence of adverse events throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.

REFERENCES:
- [Result] Aman MG, De Smedt G, Derivan A, Lyons B, Findling RL; Risperidone Disruptive Behavior Study Group. Double-blind, placebo-controlled study of risperidone for the treatment of disruptive behaviors in children with subaverage intelligence. Am J Psychiatry. 2002 Aug;159(8):1337-46. doi: 10.1176/appi.ajp.159.8.1337. PMID 12153826